CLINICAL TRIAL: NCT02018523
Title: A Pilot Study of Lenalidomide Maintenance Therapy in Stage IIIB/IV Non-small Cell Lung Cancer After First-line Chemotherapy
Brief Title: Lenalidomide Maintenance Therapy in Stage IIIB/IV Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study did not enroll enough subjects to make a statistically sound conclusion.
Sponsor: Jun Zhang (Other)
Collaborators: Celgene Corporation (Industry); Baylor College of Medicine (Other)
Responsible Party: Sponsor-Investigator, Jun Zhang, Assistant Professor, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-32774
Record Dates: First submitted 2013-12-17; First posted 2013-12-23 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Carcinoma, Non-Small-Cell Lung; Stage 3B/4; Maintenance Therapy; Lenalidomide
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide (Experimental): Oral lenalidomide 10 mg daily until disease progression
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — lenalidomide 10mg/day orally until disease progression
  Other Names: Revlimid

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of maintenance therapy with daily low dose lenalidomide in patients with stage IIIB/IV non-small cell lung cancer (NSCLC) after first line chemotherapy. Investigators expect this treatment approach will delay disease progression by boosting the patient's anti-tumor immune response. Investigators hypothesize that 10 mg/day of lenalidomide can be administered safely as maintenance therapy and improve progression free survival time.

DETAILED DESCRIPTION:
For patients with stage IIIB/IV non-small cell lung cancer, who did not progress after first line chemotherapy, lenalidomide 10mg/day orally will be administered as maintenance therapy until disease progression or death.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed stage IIIB or stage IV NSCLC with measurable disease at initial presentation prior to chemotherapy. See Section 8.4.1 for measurable disease parameters.
* Patients must have had a complete response (CR), partial response (PR) or stable disease (SD) after 4-6 cycles of first-line chemotherapy. Tumor response will be assessed by RECIST criteria version 1.1.
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, or radiotherapy before entering this study.

  1. Myelosuppressive chemotherapy: At least 21 days elapsed from end of treatment before registration (42 days if prior nitrosourea).
  2. Hematopoietic growth factors: At least 7 days since the completion of therapy with a growth factor.
  3. Other: For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur.
  4. XRT: > or = to 2 weeks for local palliative XRT (small port); 3 months must have elapsed if 50% radiation of pelvis; 6 weeks must have elapsed if other substantial bone marrow radiation.
* Patients must be > or = 18 years of age.
* ECOG performance status < or = to 1 (Karnofsky > 70%).
* Organ Functions: Patients must have normal organ and marrow function as defined below within 28 days of registration:

  1. Leukocytes > or = 3,000/uL
  2. Absolute neutrophil count > or = 1,500/uL
  3. Hemoglobin > or = 8 g/dL
  4. Platelets > or = 100,000/uL
  5. Total bilirubin 1.5X institutional upper limit of normal (ULN)
  6. AST (SGOT) and ALT (SGPT) 1.5X institutional ULN
  7. Creatinine clearance > or = 60 mL/min/1.73 m2 for patients with creatinine levels > institutional normal
* All study participants must be willing and agree to be registered into the mandatory REVLIMID REMS program, and be willing and able to comply with the requirements of REVLIMID REM. REVLIMID REMS registration does not need to be complete to determine study eligibility.
* Females of childbearing potential (FCBP)* must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days before registration. Treating investigator must affirm intention to perform another serum or urine UPT 24 hours before initiating lenalidomide treatment.

  *FCBP: A female of childbearing potential (FCBP) is a sexually mature female who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
* All patients must be counseled about pregnancy precautions, risks of fetal exposure and other risks. The counseling must be done before the initiation of the study and every 28 days before the study drug is dispensed to the subject. FCBP must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. See Appendix D: Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods.
* Able to take aspirin (81 mg) daily as prophylactic anticoagulation (Patients intolerant to ASA may use warfarin or low molecular weight heparin).
* Able to understand and willing to sign a written informed consent document.
* Life expectancy > or = 12 weeks

Exclusion Criteria

* Concomitant Medications:

  1. Patients may not be receiving any other anti-cancer therapy.
  2. Patients may not be receiving any other investigational agents.
  3. Patients may not be receiving systemic steroids or other immunosuppressive drugs; however, steroid containing inhaler may be allowed after discussing with the Principal Investigator. Duration of 5 half-lives must have elapsed before the study registration if the patient was on systemic steroids or other immunosuppressive drugs.
* Patients with untreated brain metastasis, or with treated brain metastasis but requiring steroids.
* Patients with known EGFR mutation or EML-ALK fusion gene and with stage IV disease.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to lenalidomide or thalidomide.
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, myocardial infarction within the last 6 months, unstable angina pectoris, cardiac arrhythmia, autoimmune disease or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or breastfeeding women are excluded from this study because lenalidomide has the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with lenalidomide, breastfeeding should be discontinued if the mother is treated with lenalidomide.
* Known sera-positive for or active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV). Patients who are seropositive because of hepatitis B virus vaccine are eligible.
* Any other clinically significant medical condition and/or organ dysfunction that will interfere with the administration of the therapy according to this protocol or which, in the views of investigator, preclude combination chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Progression free survival | up to 6 months from the date of registration
  Progression free survival is defined as the duration of time from the date starting lenalidomide to the date of documented radiographic progression or death.

SECONDARY OUTCOMES:
Number of participants with adverse events | From date of registration to end of study, up to 3 years
Change in circulating immune cells | Change from baseline at 1 week
Change in circulating immune cells | Change from baseline at 5 weeks
Change in circulating immune cells | Change from baseline at 9 weeks
Change in circulating immune cells | Change from baseline at 13, 17, 21 and 25 weeks
Change in circulating immune cells | Change from baseline to 6 months, 9 months and 1 year
Change in circulating immune cells | Change from baseline to 1.5, 2, 2.5 and 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, M.D., Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Background] Schiller JH, Harrington D, Belani CP, Langer C, Sandler A, Krook J, Zhu J, Johnson DH; Eastern Cooperative Oncology Group. Comparison of four chemotherapy regimens for advanced non-small-cell lung cancer. N Engl J Med. 2002 Jan 10;346(2):92-8. doi: 10.1056/NEJMoa011954. PMID 11784875
- [Background] Cappuzzo F, Ciuleanu T, Stelmakh L, Cicenas S, Szczesna A, Juhasz E, Esteban E, Molinier O, Brugger W, Melezinek I, Klingelschmitt G, Klughammer B, Giaccone G; SATURN investigators. Erlotinib as maintenance treatment in advanced non-small-cell lung cancer: a multicentre, randomised, placebo-controlled phase 3 study. Lancet Oncol. 2010 Jun;11(6):521-9. doi: 10.1016/S1470-2045(10)70112-1. Epub 2010 May 20. PMID 20493771
- [Background] Paz-Ares LG, de Marinis F, Dediu M, Thomas M, Pujol JL, Bidoli P, Molinier O, Sahoo TP, Laack E, Reck M, Corral J, Melemed S, John W, Chouaki N, Zimmermann AH, Visseren-Grul C, Gridelli C. PARAMOUNT: Final overall survival results of the phase III study of maintenance pemetrexed versus placebo immediately after induction treatment with pemetrexed plus cisplatin for advanced nonsquamous non-small-cell lung cancer. J Clin Oncol. 2013 Aug 10;31(23):2895-902. doi: 10.1200/JCO.2012.47.1102. Epub 2013 Jul 8. PMID 23835707
- [Background] Ciuleanu T, Brodowicz T, Zielinski C, Kim JH, Krzakowski M, Laack E, Wu YL, Bover I, Begbie S, Tzekova V, Cucevic B, Pereira JR, Yang SH, Madhavan J, Sugarman KP, Peterson P, John WJ, Krejcy K, Belani CP. Maintenance pemetrexed plus best supportive care versus placebo plus best supportive care for non-small-cell lung cancer: a randomised, double-blind, phase 3 study. Lancet. 2009 Oct 24;374(9699):1432-40. doi: 10.1016/S0140-6736(09)61497-5. Epub 2009 Sep 18. PMID 19767093
- [Background] Sakaguchi S, Yamaguchi T, Nomura T, Ono M. Regulatory T cells and immune tolerance. Cell. 2008 May 30;133(5):775-87. doi: 10.1016/j.cell.2008.05.009. PMID 18510923
- [Background] Al-Shibli KI, Donnem T, Al-Saad S, Persson M, Bremnes RM, Busund LT. Prognostic effect of epithelial and stromal lymphocyte infiltration in non-small cell lung cancer. Clin Cancer Res. 2008 Aug 15;14(16):5220-7. doi: 10.1158/1078-0432.CCR-08-0133. PMID 18698040
- [Background] Kawai O, Ishii G, Kubota K, Murata Y, Naito Y, Mizuno T, Aokage K, Saijo N, Nishiwaki Y, Gemma A, Kudoh S, Ochiai A. Predominant infiltration of macrophages and CD8(+) T Cells in cancer nests is a significant predictor of survival in stage IV nonsmall cell lung cancer. Cancer. 2008 Sep 15;113(6):1387-95. doi: 10.1002/cncr.23712. PMID 18671239
- [Background] Petersen RP, Campa MJ, Sperlazza J, Conlon D, Joshi MB, Harpole DH Jr, Patz EF Jr. Tumor infiltrating Foxp3+ regulatory T-cells are associated with recurrence in pathologic stage I NSCLC patients. Cancer. 2006 Dec 15;107(12):2866-72. doi: 10.1002/cncr.22282. PMID 17099880
- [Background] Shimizu K, Nakata M, Hirami Y, Yukawa T, Maeda A, Tanemoto K. Tumor-infiltrating Foxp3+ regulatory T cells are correlated with cyclooxygenase-2 expression and are associated with recurrence in resected non-small cell lung cancer. J Thorac Oncol. 2010 May;5(5):585-90. doi: 10.1097/JTO.0b013e3181d60fd7. PMID 20234320
- [Background] Erfani N, Mehrabadi SM, Ghayumi MA, Haghshenas MR, Mojtahedi Z, Ghaderi A, Amani D. Increase of regulatory T cells in metastatic stage and CTLA-4 over expression in lymphocytes of patients with non-small cell lung cancer (NSCLC). Lung Cancer. 2012 Aug;77(2):306-11. doi: 10.1016/j.lungcan.2012.04.011. Epub 2012 May 17. PMID 22608141
- [Background] Karagoz B, Bilgi O, Gumus M, Erikci AA, Sayan O, Turken O, Kandemir EG, Ozturk A, Yaylaci M. CD8+CD28- cells and CD4+CD25+ regulatory T cells in the peripheral blood of advanced stage lung cancer patients. Med Oncol. 2010 Mar;27(1):29-33. doi: 10.1007/s12032-008-9165-9. Epub 2009 Jan 16. PMID 19148592
- [Background] Elias D, Lasser PH, Desruennes E, Mankarios H, Jiang Y. Surgical approach to segment I for malignant tumors of the liver. Surg Gynecol Obstet. 1992 Jul;175(1):17-24. PMID 1621195
- [Background] Okita R, Saeki T, Takashima S, Yamaguchi Y, Toge T. CD4+CD25+ regulatory T cells in the peripheral blood of patients with breast cancer and non-small cell lung cancer. Oncol Rep. 2005 Nov;14(5):1269-73. PMID 16211295
- [Background] Woo EY, Yeh H, Chu CS, Schlienger K, Carroll RG, Riley JL, Kaiser LR, June CH. Cutting edge: Regulatory T cells from lung cancer patients directly inhibit autologous T cell proliferation. J Immunol. 2002 May 1;168(9):4272-6. doi: 10.4049/jimmunol.168.9.4272. PMID 11970966
- [Background] LeBlanc R, Hideshima T, Catley LP, Shringarpure R, Burger R, Mitsiades N, Mitsiades C, Cheema P, Chauhan D, Richardson PG, Anderson KC, Munshi NC. Immunomodulatory drug costimulates T cells via the B7-CD28 pathway. Blood. 2004 Mar 1;103(5):1787-90. doi: 10.1182/blood-2003-02-0361. Epub 2003 Sep 25. PMID 14512311
- [Background] Chang DH, Liu N, Klimek V, Hassoun H, Mazumder A, Nimer SD, Jagannath S, Dhodapkar MV. Enhancement of ligand-dependent activation of human natural killer T cells by lenalidomide: therapeutic implications. Blood. 2006 Jul 15;108(2):618-21. doi: 10.1182/blood-2005-10-4184. Epub 2006 Mar 28. PMID 16569772
- [Background] Galustian C, Meyer B, Labarthe MC, Dredge K, Klaschka D, Henry J, Todryk S, Chen R, Muller G, Stirling D, Schafer P, Bartlett JB, Dalgleish AG. The anti-cancer agents lenalidomide and pomalidomide inhibit the proliferation and function of T regulatory cells. Cancer Immunol Immunother. 2009 Jul;58(7):1033-45. doi: 10.1007/s00262-008-0620-4. Epub 2008 Nov 14. PMID 19009291
- [Background] Lu L, Payvandi F, Wu L, Zhang LH, Hariri RJ, Man HW, Chen RS, Muller GW, Hughes CC, Stirling DI, Schafer PH, Bartlett JB. The anti-cancer drug lenalidomide inhibits angiogenesis and metastasis via multiple inhibitory effects on endothelial cell function in normoxic and hypoxic conditions. Microvasc Res. 2009 Mar;77(2):78-86. doi: 10.1016/j.mvr.2008.08.003. Epub 2008 Sep 4. PMID 18805433
- [Background] Dredge K, Horsfall R, Robinson SP, Zhang LH, Lu L, Tang Y, Shirley MA, Muller G, Schafer P, Stirling D, Dalgleish AG, Bartlett JB. Orally administered lenalidomide (CC-5013) is anti-angiogenic in vivo and inhibits endothelial cell migration and Akt phosphorylation in vitro. Microvasc Res. 2005 Jan;69(1-2):56-63. doi: 10.1016/j.mvr.2005.01.002. PMID 15797261
- [Background] Eisen T, Trefzer U, Hamilton A, Hersey P, Millward M, Knight RD, Jungnelius JU, Glaspy J. Results of a multicenter, randomized, double-blind phase 2/3 study of lenalidomide in the treatment of pretreated relapsed or refractory metastatic malignant melanoma. Cancer. 2010 Jan 1;116(1):146-54. doi: 10.1002/cncr.24686. PMID 19862820
- [Background] Miller AA, Case D, Harmon M, Savage P, Lesser G, Hurd D, Melin SA. Phase I study of lenalidomide in solid tumors. J Thorac Oncol. 2007 May;2(5):445-9. doi: 10.1097/01.JTO.0000268679.33238.67. PMID 17473661
- [Background] Dahut WL, Aragon-Ching JB, Woo S, Tohnya TM, Gulley JL, Arlen PM, Wright JJ, Ventiz J, Figg WD. Phase I study of oral lenalidomide in patients with refractory metastatic cancer. J Clin Pharmacol. 2009 Jun;49(6):650-60. doi: 10.1177/0091270009335001. PMID 19451403
- [Background] Bartlett JB, Michael A, Clarke IA, Dredge K, Nicholson S, Kristeleit H, Polychronis A, Pandha H, Muller GW, Stirling DI, Zeldis J, Dalgleish AG. Phase I study to determine the safety, tolerability and immunostimulatory activity of thalidomide analogue CC-5013 in patients with metastatic malignant melanoma and other advanced cancers. Br J Cancer. 2004 Mar 8;90(5):955-61. doi: 10.1038/sj.bjc.6601579. PMID 14997189
- [Background] Sanborn SL, Gibbons J, Krishnamurthi S, Brell JM, Dowlati A, Bokar JA, Nock C, Horvath N, Bako J, Remick SC, Cooney MM. Phase I trial of docetaxel given every 3 weeks and daily lenalidomide in patients with advanced solid tumors. Invest New Drugs. 2009 Oct;27(5):453-60. doi: 10.1007/s10637-008-9200-x. Epub 2008 Nov 15. PMID 19011760
- [Background] Kalmadi S, Davis M, Dowlati A, O'Keefe S, Cline-Burkhardt M, Pelley RJ, Borden E, Dreicer R, Bukowski R, Mekhail T. Phase I trial of three-weekly docetaxel, carboplatin and oral lenalidomide (Revlimid) in patients with advanced solid tumors. Invest New Drugs. 2007 Jun;25(3):211-6. doi: 10.1007/s10637-006-9025-4. Epub 2006 Nov 11. PMID 17103043
- [Background] Attal M, Lauwers-Cances V, Marit G, Caillot D, Moreau P, Facon T, Stoppa AM, Hulin C, Benboubker L, Garderet L, Decaux O, Leyvraz S, Vekemans MC, Voillat L, Michallet M, Pegourie B, Dumontet C, Roussel M, Leleu X, Mathiot C, Payen C, Avet-Loiseau H, Harousseau JL; IFM Investigators. Lenalidomide maintenance after stem-cell transplantation for multiple myeloma. N Engl J Med. 2012 May 10;366(19):1782-91. doi: 10.1056/NEJMoa1114138. PMID 22571202
- [Background] McCarthy PL, Owzar K, Hofmeister CC, Hurd DD, Hassoun H, Richardson PG, Giralt S, Stadtmauer EA, Weisdorf DJ, Vij R, Moreb JS, Callander NS, Van Besien K, Gentile T, Isola L, Maziarz RT, Gabriel DA, Bashey A, Landau H, Martin T, Qazilbash MH, Levitan D, McClune B, Schlossman R, Hars V, Postiglione J, Jiang C, Bennett E, Barry S, Bressler L, Kelly M, Seiler M, Rosenbaum C, Hari P, Pasquini MC, Horowitz MM, Shea TC, Devine SM, Anderson KC, Linker C. Lenalidomide after stem-cell transplantation for multiple myeloma. N Engl J Med. 2012 May 10;366(19):1770-81. doi: 10.1056/NEJMoa1114083. PMID 22571201